CLINICAL TRIAL: NCT02438579
Title: Edinburgh and Lothians Viral Intervention Study (ELVIS). A Pilot Randomised Control Trial of Hypertonic Saline Nasal Irrigation and Gargling on Individuals With the Common Cold to Assess Recruitment, Retention, Side Effects & Effectiveness
Brief Title: Hypertonic Saline Nasal Irrigation and Gargling for the Common Cold.
Acronym: ELVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Collaborators: University of Edinburgh (Other)
Responsible Party: Principal Investigator, Dr. Sandeep Ramalingam, Consultant Virologist, NHS Lothian
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13/SS/0079; 10-303 (Other Grant/Funding Number: Edinburgh & Lothians Health Foundation)
Record Dates: First submitted 2015-02-16; First posted 2015-05-08 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Common Cold; Upper Respiratory Tract Infections
Keywords: Hypertonic saline; nasal irrigation; gargling; URTI
MeSH Terms: conditions — Common Cold; Respiratory Tract Infections | interventions — Nasal Lavage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Irrigation & Gargling (Experimental): Videos on how to collect nasal swabs, prepare and perform hypertonic saline nasal irrigation and gargling (HSNIG) are shown. A nasal swab is collected. Participant chooses the highest concentration of hypertonic saline he/she is comfortable with (from 1.5, 2.0, 2.5 and 3.0%) and performs HSNIG under observation. Nasal swabs are to be collected first thing in the morning on 4 consecutive days and posted using the Royal Mail Safebox. Daily diaries are to be completed (online / paper form) until they document "not unwell" for two consecutive days; or a maximum of 14 days or if they need medical attention for the URTI. Swabs are tested in parallel to detect change in viral shedding.
  Interventions: Other: Nasal Irrigation & Gargling
- Control (No Intervention): The control group are advised to manage the URTI as they normally do. A video on how to collect nasal swabs is shown. A nasal swab is collected. Nasal swabs are to be collected first thing in the morning on 4 consecutive days and posted using the Royal Mail Safebox. Daily diaries are to be completed (online / paper form) until they document "not unwell" for two consecutive days; or a maximum of 14 days or if they need medical attention for the URTI. Swabs are tested in parallel to detect change in viral shedding.

INTERVENTIONS:
Other: Nasal Irrigation & Gargling — Participants are advised to perform the intervention as frequently as required (expected frequency around 6 times a day for the first two days, reducing in frequency from day 3 as symptoms improve).
  Arms: Nasal Irrigation & Gargling

SUMMARY:
Viral upper respiratory tract infections (URTI), one of the commonest infection faced by humans, have a significant impact on individuals, families, health service and economy. Though rhinoviruses are called the "common cold virus", numerous viruses can cause URTI. Hence virus specific remedy for URTI is impractical. There are currently no evidence-based interventions that reduce the severity, symptom duration or viral shedding. Preliminary evidence suggests that hypertonic saline nasal irrigation and gargling (HSNIG) may reduce the duration of symptoms.

With this pilot randomised controlled trial (RCT), the investigators aim to assess the feasibility of undertaking a definitive RCT of HSNIG in adults with URTI. This pilot focuses on recruitment rate, willingness to be randomised, acceptability, compliance and likely effect size of the intervention.

This pilot RCT compares HSNIG vs. usual care in 60 adults. Serial self-collected mid-turbinate swabs will help assess change in viral shedding. Symptomatic relief is measured by a validated symptom score. A questionnaire based participant feedback will help assess intervention and trial procedures.

This mixed-methods pilot trial will help inform plans for a definitive RCT of this low-cost intervention that has the potential of substantial health and societal benefits.

DETAILED DESCRIPTION:
1. Aims:

   To assess the feasibility of undertaking a RCT of HSNIG in adults with URTI focusing on recruitment rate, willingness to be randomised, acceptability, compliance and likely effect size of the intervention.

   1.1. Research questions:
   1. What is the likely rate of recruitment and loss to follow-up?
   2. Are the study procedures acceptable to participants?
   3. Is there a likely reduction in duration of symptoms and viral shedding?
   4. What effect size is estimated for the definitive trial in relation to duration of symptoms and improvement in quality-of-life?
2. Subjects:

   2.1 Sample size: This is a pilot trial so no formal sample size calculations are indicated. However, with a sample size of 27 per group the investigators would be able to express the proportion of those who return the symptom score diary and samples within that group to within ±19% based on a two-sided 95% confidence interval around an expected proportion of 0.5. With the two groups combined [i.e. a sample size of 54] the investigators would be able to express a proportion to within ±13%. To allow for 10% dropouts the sample size has been increased to 30 per group.

   2.2 Recruitment: The investigators propose to enrol a total of 60 participants (30/arm) for this pilot. The investigators plan to recruit by advertising the study in the community by the following routes.
   * Sending flyers to parents through schools run by Edinburgh and Midlothian councils.
   * Study website (www.elvisstudy.com), National Health Service (NHS) Lothian, University of Edinburgh websites.
   * Local media coverage by way of interviews.
   * Flyers in workplaces with large numbers of staff (e.g. banks, supermarkets, councils).
   * Posters in pharmacies and General practitioner (GP) surgeries.

   Interested individuals will be asked to contact the trial nurse at the clinical research facility (CRF) situated at the Royal Infirmary of Edinburgh (RIE) and Western General Hospital within 48 hours of symptom onset. The trial nurse will consent, randomise, and recruit volunteers. Participants will be advised to go to their GP as per norm if they become unwell and that they can withdraw from the study if they so wish for other reasons. At the end of their participation in the study, they will be given £30 as recompense for any inconvenience.
3. Research Methods:

   3.1 Randomisation: Participants are randomised in a 1:1 ratio to receive intervention or control, this has been done using an online randomisation minimised by sex (M/F) and smoking status (current/not a current smoker) and allocated to each treatment arm with a probability 0.9 to ensure a random allocation.

   3.2 Instructions to participants: 3.2.1 Both arms: Participants are taught to complete (online or paper) a modified short Wisconsin upper respiratory symptom survey (WURSS-21-Scot) and the EQ-5D-5L questionnaire. Baseline symptom scores are recorded by the participant.

   Participants are taught to collect nasal swabs. A baseline swab is collected under observation and sent to the virology laboratory at the Royal Infirmary of Edinburgh (RIE). Swabs, transport medium and Royal Mail Safebox will be provided to the participant to collect a nasal swab first thing in the morning (before HSNIG for the intervention arm) for four consecutive days and return to the laboratory.

   3.2.2 Intervention arm: The intervention group will be shown a video on preparing the hypertonic sea-salt solution and how to perform HSNIG. They will be asked to perform the procedure under supervision. The trial nurse will help them identify the highest concentration of saline they are comfortable with. Participants are advised to perform the intervention as frequently as required (expected frequency around 6 times/day for the first two days, reducing in frequency from day 3 as symptoms improve). A package containing instructions, digital-measuring spoon, sea-salt, and equipment for irrigation and flask (if they wish to prepare solution for multiple uses during the day) will then be handed over to the participant. Participants in the intervention arm will also document compliance and side effects daily

   3.2.3 Control arm: They are advised to manage the URTI as they normally do.

   3.3 Data collection: 3.3.1 "WURSS-21-Scot" diary and EQ-5D-5L Questionnaire: All participants will complete the "WURSS-21-Scot" diary at a set time during the day. Participants will answer the question "how unwell do you feel today". If they score >0, then symptoms and functional ability are graded 0-7. They then answer the global change question. Total score/day is calculated by summing the scores of all 10 symptoms daily. All participants will also answer the EQ-5D-5L questionnaire.

   The following information is collected at recruitment: where they heard about the study, influenza vaccination history, number of family members and whether sufficient information was provided.

   The intervention arm will also answer the following questions daily: how many times they performed HSNIG, if they performed one or both parts of HSNIG and if there were any side effects.

   Both arms will answer if they had to take any medications for the URTI and whether they needed to contact the GP for further management of their URTI.

   Diaries are maintained until participant records "not unwell" on two consecutive days or for a maximum of 14 days or until follow up is terminated because the individual needs further treatment.

   3.3.2 Virology: Swabs will be sent to the Department of Virology, RIE for testing. Baseline samples will be tested to identify individuals in whom an aetiology can be proven. If a viral aetiology is identified, all samples (day 0 - day 4) will be tested in parallel to identify change in viral shedding.

   3.3.3 Data collection procedures: The trial nurse will follow up participants who do not complete the diary or return samples (after 48 hours of expected return). Information on number of family members with URTI will be collected at the end of the study. Feedback will be collected from participants after the follow-up period. These will address acceptability, health service use, costs to the patient and suggestions for improving the study procedures for the main trial.
4. Data Analysis:

The number of participants returning swabs, completing diaries and following treatment as per protocol will be presented as percentages (with 95% confidence intervals). The investigators will present recruitment as an overall rate, but also graphically as there is likely to be seasonal variation. Using results from the swabs the investigators will determine when a person stops viral shedding and, using chi-square and chi-square test for trend, determine if there is a relationship between groups. Using two-sample t-tests or non-parametric equivalent as appropriate the investigators will determine if there is any evidence of a difference in the duration of symptoms and symptom severity [as defined by the maximum WURSS-21-Scot score over treatment period]. Feedback will be analysed using a conventional content analysis approach, with emerging findings discussed by the research team to aid interpretation of findings.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of upper respiratory tract infection (URTI)
* Within 48 hours of onset

Exclusion Criteria:

* Onset of URTI >48 hours
* On antibiotics
* Pregnancy
* History of chronic illness or immunosuppression
* Allergic rhinitis
* Unable to perform nasal irrigation and gargling
* Taking part in another medical trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
What is the recruitment rate? | 6 months
  A standard accrual plot will be produced, a plot of number of participants recruited in each week and the recruitment rate will be expressed as the average number of participants recruited per week over the duration of the study period. A table showing number of participants recruited by site will also be produced.

SECONDARY OUTCOMES:
What is the rate of sample return within the two arms? | 6 months
  The overall number of participants returning swabs, will be presented as numbers/percentages [with 95% confidence intervals (CI) for the percentages]. Differences between the groups will be assessed using a binomial test for the comparison of proportions and expresses as a percentage [with 95% CI].
What is the rate of diary completion within the two arms? | 6 months
  The overall number of participants completing diaries will be presented as numbers/percentages [with 95% CI]. Differences between the groups will be assessed using a binomial test for the comparison of proportions and expresses as a percentage [with 95% CI].
Do the participants comply with the intervention regime? | 6 months
  The overall number of participants following treatment as per protocol will be presented as numbers/percentages [with 95% CI]. Differences between the groups will be assessed using a binomial test for the comparison of proportions and expresses as a percentage [with 95% CI].
What are the participant views on acceptability? | 6 months
  Responses to participant acceptability will be presented as numbers and percentages split by treatment arm.
Is there a difference between arms in their quality-of-life? | 6 months
  A persons average quality of life as measured by the EQ-VAS daily over the study period will be calculated and compared between treatment groups using a two-sample t-test or non-parametric equivalent as appropriate. Rate of change will also be compared between groups in the same manner where the rate of change will be determined by: ([final day EQ-VAS] - [baseline EQ-VAS]) / (number of days - 1)
Is there a difference between arms in the duration of symptoms or viral shedding? | 6 months
  Duration of symptoms will be defined by WURSS-21-Scot [time to reach a score of 0 for two consecutive days]. If appropriate to treat as a continuous variable, a two-sample t-test or non-parametric equivalent will be used as appropriate. However it may be more appropriate to treat the time a categorical measure, if this is the case we will use Chi-square/Chi-square test for trend as appropriate. In addition to this the average WURSS-21-Scot will be compared between treatment arms using the same methods.
  Chi-square test and chi-square test for trend will be used as appropriate to determine if there is a difference in viral shedding between arms. Viral load is measured daily for the first 4 days and reported using CT values, we will estimate the slope of the line for each participant and a comparison will be made between groups. In addition to this average CT value and average log copies above level of detection will be compared across groups using a two-sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Ramalingam, PhD, FRCPath, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Background] Barrett B, Brown RL, Mundt MP, Thomas GR, Barlow SK, Highstrom AD, Bahrainian M. Validation of a short form Wisconsin Upper Respiratory Symptom Survey (WURSS-21). Health Qual Life Outcomes. 2009 Aug 12;7:76. doi: 10.1186/1477-7525-7-76. PMID 19674476